CLINICAL TRIAL: NCT06404541
Title: A Comparison Between the Ocular Surface of Different Concentrations of Benzalkonium Chloride Preservative in Postoperative Topical Medications After Cataract Surgery
Brief Title: A Comparative Study Between Preservative With Benzalkonium Chloride vs Preservative Free Eye Drops on the Ocular Surface
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, Amnah Ayman, AAyman, Kasr El Aini Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MS-127-2023
Record Dates: First submitted 2024-05-05; First posted 2024-05-08 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Ocular Surface Disease; Dry Eye Syndromes
MeSH Terms: conditions — Dry Eye Syndromes | interventions — Dexamethasone; Tobramycin

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A (Active Comparator): 20 eyes received single dose unit Dexathalm containing: actives: In 1ml: Dexamethason 1mg and Netilimicin 3mg, without preservatives 5 times per day.
  Interventions: Drug: Dexamethasone, tobramycin, netilimicin
- Group B (Active Comparator): 20 eyes received regular Tobradex eye drops containing actives: In 1 ml: tobramycin 3 mg and dexamethasone 1 mg, preservative: 0.1mg of BAK per ml 5 times per day.
  Interventions: Drug: Dexamethasone, tobramycin, netilimicin
- Group C (Active Comparator): 20 eyes received Dexathalm multi-dose containing actives: In 1ml: Dexamethasone 1mg and Netilimicin 3mg, preservatives: 0.05mg of BAK per ml 5 times per day.
  Interventions: Drug: Dexamethasone, tobramycin, netilimicin

INTERVENTIONS:
Drug: Dexamethasone, tobramycin, netilimicin — Group A: Dexathalm single dose Group B: Tobradex Group C: Dexathalm multi-dose

SUMMARY:
study the effect of different concentrations of benzalkonium chloride on the ocular surface of non-dry-eyed patients post cataract surgery.

DETAILED DESCRIPTION:
60 eyes of will be included in this study.

* 20 eyes will receive regular Tobradex 0.1mg/ml BAK 5 times per day (Group 1).
* 20 eyes will receive Dexathalm multidose 0.05mg/ml BAK 5 times per day (Group 2).
* 20 eyes will receive single dose unit Dexathalm NO BAK 5 times per day (Group 3).

Preoperative assessment:

All selected patients will receive thorough explanation of the study design and aims, an informed consent will be obtained from all patients.

Tear break up time (TBUT) will be measured non-invasively by Ocular Surface analyzer.

Ocular Surface disease index will be calculated by filling a questionnaire. 12-item questionnaire provide a rapid assessment of the symptoms of ocular irritation consistent with dry eye disease and their impact on vision-related functioning.

Postoperative:

1. All patients will be examined at day1, 1 week and 3 week postoperative.
2. At 3 weeks re-evaluate I. TBUT by non-invasive ocular surface analyzer II. OSDI by filling the questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing uncomplicated cataract surgery
* Cataract grade: (LOCSIII): NO2NC2,C3,P2

Exclusion Criteria:

Preoperative non-invasive TBUT<10 seconds. Patients who have rheumatoid arthritis or autoimmune diseases affecting corneal surface.

Involutional entropion or ectropion preoperative Postoperative significant corneal edema requiring medication.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-01-10 (Actual); Primary Completion 2024-04-10 (Actual); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
NBUT | preoperative and 1 month postoperative
  non invasive tear break up time
TMH | preoperative and 1 month postoperative
  Tear meniscus Height
OSDI | preoperative and 1 month postoperative
  ocular surface disease index
MG loss | preoperative and 1 month postoperative
  meibomian gland loss

CONTACTS AND LOCATIONS:
Locations (1):
- KasrAl Ainy Hospital, Cairo, Giza Governorate, Egypt